CLINICAL TRIAL: NCT04632823
Title: "The Effect of Comprehensive Non-pharmacological Treatment on Metabolic Disorders in Type 2 Diabetic Patients"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Astana Medical University (Other)
Responsible Party: Principal Investigator, Viktoriya Li, PhD, Head of Rehabilitation, Astana Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AstanaMU-1
Record Dates: First submitted 2020-11-09; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes mellitus; non-pharmacological treatment; lifestyle intervention; structured program
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: prospective, single-center
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive non-pharmacological program intervention (Experimental): The experimental group receives usual diabetes care plus 24 weeks of the comprehensive non-pharmacological program intervention.
  Interventions: Combination Product: Comprehensive Non-pharmacological Treatment Program
- Usual diabetes care (No Intervention): This group is control, the patients receive usual diabetes care routines.

INTERVENTIONS:
Combination Product: Comprehensive Non-pharmacological Treatment Program — dietary supplement, specific type of exercise, self-management education
  Arms: Comprehensive non-pharmacological program intervention

SUMMARY:
Evaluation of the effectiveness of comprehensive non-pharmacological treatment on metabolic disorders in type 2 diabetic patients

DETAILED DESCRIPTION:
Patients in the intervention group will participate in a comprehensive non-pharmacological treatment of type 2 diabetes, the main components are:

* changing the meal plan (individual and group counseling, assistance in developing menus and determining the calorie intake, keeping a food diary)
* individually dosed physical exercises using specific exercise program;
* comprehensive training (course of interactive lessons, self-control training). The program included group sessions with a team of specialists: nutritionist, endocrinologist, physical therapy doctor and included 3 sessions per week for 24 weeks. Each visit included teaching patients in a group format and in an interactive form (classes with specialists alternated), performing physical exercises using the specific exercise program under the supervision of a physiotherapy physician, evaluating medical indicators, and a self-control diary.

Patients in the control group will not participate in group sessions, but they had the opportunity to receive non-pharmacological care provided in the framework of free outpatient care. Their indicators will be recorded during a routine visit to the doctor at the baseline, after 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* medically diagnosed with type 2 diabetes mellitus
* HbA1c result of ≤7.0% within the past 2 months
* body mass index (BMI) of ≥26 kg/m^2
* hypoglycemic therapy: metformin only

Exclusion Criteria:

* pregnancy
* the use of other hypoglycemic drugs
* the use of medication for weight loss
* cardiovascular diseases (heart attack or cardiac procedure within the past 3 months)
* had stroke or history of treatment for transient ischemic attacks in the past 3 months
* had chronic renal failure or were on dialysis
* any conditions that do not allow the patient to perform the complex of the proposed physical exercises

Ages: 45 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Glycosylated Hemoglobin at 6 months | at baseline and at 24-week postrandomization
  HbA1c value
Change from Baseline Body Mass Index at 6 months | at baseline and at 24-week postrandomization
  BMI

SECONDARY OUTCOMES:
Change from Baseline Blood Pressure at 6 months | at baseline and at 24-week postrandomization
  Systolic and diastolic blood pressure at the brachial artery
Change from Baseline Lipid Profiles at 6 months | at baseline and at 24-week postrandomization
  Total Triglyceride, Total Cholesterol, high-density lipoprotein (HDL), and low-density lipoprotein (LDL)
Change from Baseline Homeostasis ModelAssessment of Insulin Resistance at 6 months (HOMA-IR) | at baseline and at 24-week postrandomization
  Homeostasis ModelAssessment of Insulin Resistance

CONTACTS AND LOCATIONS:
Overall Officials: Viktoriya Li, PhD, Principal Investigator — Astana Medical University
Locations (4):
- Kazakhstan (3):
  - West Kazakhstan Marat Ospanov Medical University, Aktobe, Aktobe Region
  - Astana Medical University, Astana
  - The Center for Preventive Medicine and Life Extension of Nur-Sultan, Astana
- National Medical Research Center for Endocrinology, Ministry of Health of the Russian Federation, Moscow, Russia